CLINICAL TRIAL: NCT00135096
Title: APIDRA® (Insulin Glulisine) Administered Premeal vs Postmeal in Adult Subjects With Type 2 Diabetes Mellitus Receiving LANTUS® (Insulin Glargine) as Basal Insulin: a Multicenter, Randomized, Parallel, Open Label Clinical Study
Brief Title: Insulin Glulisine Administered Pre-meal Versus Post-meal in Adult Subjects With Type 2 Diabetes Mellitus Receiving Insulin Glargine as Basal Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3503
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine; Insulin Glargine

ARMS (2):
- 1 (Experimental): PREMEAL ARM: Subjects randomized to this arm will receive Apidra administered three times per day 0-15 min before the three main meals; metformin (if applicable); and Lantus qd for 52 weeks.
  Interventions: Drug: insulin glulisine
- 2 (Experimental): POSTMEAL ARM: Subjects randomized to this arm will receive Apidra administered three times per day immediately after a meal (20 min after the start of a meal); metformin (if applicable); and Lantus qd for 52 weeks.
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin glulisine — PREMEAL ARM: Subjects randomized to this arm will receive Apidra administered three times per day 0-15 min before the three main meals; metformin (if applicable); and Lantus qd for 52 weeks.
  Arms: 1
Drug: insulin glargine — POSTMEAL ARM: Subjects randomized to this arm will receive Apidra administered three times per day immediately after a meal (20 min after the start of a meal); metformin (if applicable); and Lantus qd for 52 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the change in weight from baseline to study week 52 in the per-protocol population of pre-meal insulin glulisine (Apidra) versus post-meal Apidra, in patients receiving insulin glargine (Lantus) as basal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus for at least six months
* 18 to 70 years of age, inclusive
* A1c ≥ 7.5% and ≤ 10%
* At least 3 months of continuous insulin and/or insulin analogue therapy (on at least 2 injections per day) +/- metformin prior to study entry
* Negative glutamic acid decarboxylase (GAD) autoantibodies
* Ability and willingness to perform self-monitoring of blood glucose (SMBG) at least four times a day, and at least 7 times daily during the 7-point blood glucose (BG) profile measurement days
* Ability and willingness to adhere to, and be compliant with, the study protocol
* Must be able to read English or Spanish at the sixth grade level in order to complete the patient-reported outcomes component of the study
* Signed informed consent

Exclusion Criteria:

* Subjects treated with sulfonylureas, thiazolidinediones (TZDs), or any other oral antidiabetic drugs (at study entry) except for insulin and/or insulin analogues with or without metformin
* Planned pregnancy; or pregnant or lactating females
* For subjects treated with metformin: serum creatinine ≥ 1.5 mg/dL (133 µmol/L) for males or ≥ 1.4 mg/dL (124 µmol/L) for females
* Serum creatinine ≥ 3.0 mg/dL (266 µmol/L)
* Any clinically significant renal disease (other than proteinuria) or hepatic disease
* Serum ALT or AST levels greater than 2.5 X the upper limit of normal
* Any current malignancy or any cancer within the past 5 years (except for adequately treated basal cell skin cancer or cervical carcinoma in situ)
* Diagnosis of dementia or mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Diagnosis of impaired dexterity or vision rendering the subject unable to administer multiple daily injections (MDIs)
* Cardiac status New York Heart Association (NYHA) III-IV
* Hypersensitivity to Lantus or Apidra or any of their components
* Any disease or condition (including abuse of illicit drugs, prescription medicines or alcohol) that, in the opinion of the investigator or sponsor, may interfere with the completion of the study.
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2004-08; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Compare change in weight from baseline to study week 52 in the per-protocol population of premeal Apidra vs postmeal Apidra, in patients receiving Lantus as basal insulin | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barch, B.S., Study Director — Sanofi
Locations (1):
- Sanofi-aventis, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Ratner R, Wynne A, Nakhle S, Brusco O, Vlajnic A, Rendell M. Influence of preprandial vs. postprandial insulin glulisine on weight and glycaemic control in patients initiating basal-bolus regimen for type 2 diabetes: a multicenter, randomized, parallel, open-label study (NCT00135096). Diabetes Obes Metab. 2011 Dec;13(12):1142-8. doi: 10.1111/j.1463-1326.2011.01478.x. PMID 21812890